CLINICAL TRIAL: NCT05371860
Title: Radiation Omission in Patients With HER2 Overexpressing Tumors With Pathologic
Brief Title: Radiation Omission in Patients With HER2 Overexpressing Tumors With Pathologic Complete Response
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI voluntarily closed the study. Will be reopened as a national cooperative group trial.
Sponsor: Armando Giuliano (Other)
Responsible Party: Sponsor-Investigator, Armando Giuliano, Chief, Surgical Oncology, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021-10-Giuliano-OmitRT
Record Dates: First submitted 2022-04-20; First posted 2022-05-12 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
Keywords: HER2; partial mastectomy; lumpectomy; sentinel node biopsy; axillary node dissection; pathologic complete response; breast cancer; HER2-positive
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omit breast radiation (Experimental)
  Interventions: Other: Omit breast radiation

INTERVENTIONS:
Other: Omit breast radiation — Omit breast radiation for 3 years after surgery

SUMMARY:
The purpose of this study is to evaluate the feasibility, based on recruitment rate over a 3-year period, of enrolling patients for the omission of post-operative breast radiation following breast conserving surgery and sentinel node biopsy or axillary lymph node dissection in women with HER2+ breast cancer who achieve pathologic complete response.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 40 years
* Patients must have a tissue diagnosis of HER2+ breast cancer
* Patients must have documented clinical T1-3, N0, M0 disease prior to receiving neo-adjuvant chemotherapy
* Patients must have undergone neo-adjuvant chemotherapy and targeted HER2 therapy prior to surgery and plan for completion of adjuvant systemic therapy as directed by their medical oncologist
* Patients must have completed partial mastectomy/lumpectomy and sentinel node biopsy or axillary node dissection.
* Patient must have documented pathologic complete response (defined as no residual invasive or in situ disease in the breast or axilla, including free of isolated tumor cells or micrometastasis)

Exclusion Criteria:

* Breastfeeding
* Prior history of breast cancer (invasive or ductal carcinoma in-situ) in either breast
* Prior adjuvant radiation therapy
* Patients with diagnosis of inflammatory breast cancer
* Patients with known BRCA mutation or other known breast cancer related deleterious mutations

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrolling patients measured by proportion of recruited patients to participate in the trial | At time of consent. Assessed up to 3 years
  Measured by the number of recruited patients over the number of patients approached to participate to the trial. Feasibility will be defined as recruitment rate of greater or equal to 25% among patients who are eligible to participate in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Armando Giuliano, MD, FACS, FRCSEd, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States